CLINICAL TRIAL: NCT07151677
Title: Pre-Frontal tDCS as a Novel Intervention to Reduce Effects of Post-Stroke Fatigue While Improving Language and Attention in Aphasia
Brief Title: Brain Stimulation Effects on Post-Stroke Fatigue and Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Syracuse University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DC021677-01A1 (NIH); 1R01DC021677-01A1 (NIH)
Record Dates: First submitted 2025-08-18; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Aphasia Following Cerebral Infarction; Stroke Ischemic; Fatigue Symptom
Keywords: aphasia; fatigue; post-stroke fatigue; tDCS; brain stimulation; language treatment; language therapy; speech therapy; speech-language therapy
MeSH Terms: conditions — Ischemic Stroke; Fatigue; Aphasia; Communication Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (4):
- active tDCS plus attention-focused language treatment (Experimental): active tDCS and attention focused language treatment will be administered
  Interventions: Device: tDCS (active); Behavioral: Attention-focused sentence comprehension treatment
- active tDCS plus sentence picture matching treatment (Active Comparator): active tDCS and sentence picture matching treatment will be administered
  Interventions: Device: tDCS (active); Behavioral: Sentence comprehension treatment
- sham tDCS plus attention-focused language treatment (Sham Comparator): sham tDCS and attention focused language treatment will be administered
  Interventions: Behavioral: Attention-focused sentence comprehension treatment; Device: tDCS (sham)
- sham tDCS plus sentence picture matching treatment (Sham Comparator): sham tDCS and sentence picture matching treatment will be administered
  Interventions: Behavioral: Sentence comprehension treatment; Device: tDCS (sham)

INTERVENTIONS:
Device: tDCS (active) — The investigators will administer active tDCS to left dorsolateral prefrontal cortex (DLPFC) during 10 sessions of behavioral treatment. For active tDCS, the current will slowly be increased to 2mA and applied for 20 minutes.
  Other Names: transcranial direct current stimulation
  Arms: active tDCS plus attention-focused language treatment; active tDCS plus sentence picture matching treatment
Behavioral: Attention-focused sentence comprehension treatment — This is a specific type of speech-language therapy that focuses on simultaneously improving auditory comprehension and behavioral attention. Participants will receive 10 sessions of this treatment.
  Arms: active tDCS plus attention-focused language treatment; sham tDCS plus attention-focused language treatment
Behavioral: Sentence comprehension treatment — This is a specific type of speech-language therapy that focuses on improving auditory comprehension . Participants will receive 10 sessions of this treatment.
  Arms: active tDCS plus sentence picture matching treatment; sham tDCS plus sentence picture matching treatment
Device: tDCS (sham) — The investigators will administer sham tDCS to left dorsolateral prefrontal cortex (DLPFC) during 10 sessions of behavioral treatment. For sham tDCS, the current will slowly be increased to 2mA over the course of 30 seconds and then immediately ramped back down to zero.
  Other Names: transcranial direct current stimulation
  Arms: sham tDCS plus attention-focused language treatment; sham tDCS plus sentence picture matching treatment

SUMMARY:
The goal of this clinical trial is to determine if electrical brain stimulation applied to the front parts of the brain can help people who have had a stroke improve their fatigue, language, and attention. The main question it aims to answer is:

* Does transcranial direct current stimulation (tDCS) administered to the pre-frontal areas of the brain improve post-stroke fatigue and aphasia?
* What kinds of participant characteristics are associated with better improvement of post-stroke fatigue and aphasia?

Researchers will compare active electrical stimulation to sham stimulation to see if the active stimulation does a better job at reducing fatigue and language deficits after stroke. Participants will be asked to complete fatigue, language, and cognitive testing before and after receiving 10 sessions of tDCS plus speech and language therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. No diagnosis of neurological disorder (other than stroke).
3. No diagnosis of psychiatric disorder, with the exception of anxiety and/or depression if it is managed through medication and/or behavioral intervention.
4. No seizure within the past 6 months.
5. Not pregnant.
6. Does not currently have cardiac pacemaker
7. In chronic phase of recovery, defined as at least 6 months post-stroke.
8. Not undergoing speech and language therapy targeting auditory comprehension or attention for the duration of the study.
9. No metal implants in the scalp or bone in the pre-frontal area of the head.
10. No unhealed skull fractures.
11. Onset of aphasia related to single, left hemisphere, ischemic stroke.
12. Damaged brain tissue from stroke does not overlap with left hemisphere dorsolateral prefrontal cortex.
13. Mild to moderate aphasia (as measured by WAB-R **or QAB).
14. Self-report of post-stroke fatigue (as measured on SF-CAT)
15. No significant challenges with vision or hearing (with use of corrective aids if needed; eyeglasses, hearing aids).
16. Willing to allow audio-recording of study sessions.

Exclusion Criteria:

1. Younger than 18 years old.
2. Diagnosis or history of neurological disorder other than stroke.
3. Diagnosis or history of psychiatric disorder with the exception of anxiety and/or depression if it is managed through medication and/or behavioral intervention.
4. History of seizures within the past 6 months.
5. Pregnant.
6. Currently has cardiac pacemaker
7. <6 months post-stroke (however, if this is only exclusionary criterion met, participant can be re-evaluated at the 6-month mark if still interested in the study)
8. Currently undergoing speech and language therapy targeting auditory comprehension or attention.
9. Metal implants in the scalp or bone in the pre-frontal area of the head.
10. Currently has an unhealed skull fracture.
11. Onset of aphasia related to etiology other than ischemic left hemisphere stroke.
12. Damaged brain tissue significantly overlaps with left hemisphere dorsolateral prefrontal cortex.
13. No aphasia or severe aphasia (as measured by WAB-R **or QAB).
14. Does not report experience of post-stroke fatigue (as measured on SF-CAT)
15. Significant challenges with vision and/or hearing (even with use of corrective aids).
16. Unwilling to allow audio-recording of study sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Fatigue Interference and Severity Scale for Aphasia (FISS-A) | baseline; within 1 week following the final treatment session; 3- month follow-up
  Scale from 1-7, higher scores mean more significant fatigue

SECONDARY OUTCOMES:
Continuous Performance Test (CPT) | baseline; within 1 week following the final treatment session; 3- month follow-up
Attention Network Test (ANT) | baseline; within 1 week following the final treatment session; 3- month follow-up
Sentence comprehension task | baseline; within 1 week following the final treatment session; 3- month follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Syracuse University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Yes
Data generated for this project will include participant demographic data, medical information related to the participant's stroke (e.g., date of stroke onset, lesion location), standardized test scores from language and cognitive tests (e.g., Western Aphasia Battery), and outcome measure data. All data will be de-identified.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Shared data and supporting information generated from this project will be made available as soon as possible, and no later than one year following the end of the funding period (11/30/2029). The duration of preservation and sharing of the data will be a minimum of 6 years after the end of the funding period.
Access Criteria: Controlled access will not be used. The data that is shared will be shared by unrestricted download. All datasets that can be shared will be deposited in Open Science Framework. Open Science Framework provides searchable study-level metadata for dataset discovery. Open Science Framework assigns DOIs as persistent identifiers and has a robust preservation plan to ensure long-term access. Data will be discoverable online through standard web search of the study-level metadata as well as the persistent pointer from the DOI to the dataset.
URL: https://doi.org/10.48321/D17S7Q